CLINICAL TRIAL: NCT02365792
Title: Efficacy of a Clinical Decision Support System in Prehospital Care: Single Blind, Randomized Clinical Trial.
Brief Title: Professional Development in Emergency Medical Services
Acronym: ProDEms
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Olivier Hoogmartens, Head of the Academic Center for General Practice, KU Leuven
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: ProDEmsTrial
Record Dates: First submitted 2014-06-21; First posted 2015-02-19 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Clinical Decision Support; Clinical Practice Guidelines; Emergency Medical Services
Keywords: Clinical Decision Support; Clinical Practice Guidelines; Emergency Medical Services

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CDSS1 (Active Comparator): The CDSS1 will provide decision support according to existing protocols for clinical procedures and medical treatment, mainly starting from specific symptoms or diagnostic related patients groups. The symptom oriented approach is categorised in a specific list of predetermined conditions.
  Interventions: Procedure: Clinical Decision Support Tool for Prehospital Care
- CDSS2 (Active Comparator): The CDSS2 will provide decision support according to existing protocols for clinical procedures and medical treatment, mainly starting from specific symptoms or diagnostic related patients groups. The symptom oriented approach is categorised in a specific list of predetermined conditions.
  Interventions: Procedure: Clinical Decision Support Tool for Prehospital Care
- Booklet (Placebo Comparator): The control group will provide prehospital patient care with usual decision support: a pocket-size booklet, backed by a mobile phone through which the PIT can get in contact with an Emergency Physician.
  Interventions: Procedure: Clinical Decision Support Tool for Prehospital Care

INTERVENTIONS:
Procedure: Clinical Decision Support Tool for Prehospital Care — A clinical decision support system (CDSS) is a health information technology system that is designed to assist physicians and other health professionals with clinical decision-making tasks. A working definition of the Centre for Health Evidence: "Clinical Decision Support systems link health observations with health knowledge to influence health choices by clinicians for improved health care".
  Other Names: CDSS

SUMMARY:
The ProDEms-trial focuses on nurses and ambulance drivers working in prehospital care, taking care on the one hand of patients suffering from time-sensitive critical conditions like STEMI, acute stroke or severe traumatic brain injury, and on the other hand of patients whose lives are not in immediate danger but suffer from acute exacerbation of chronic conditions or suffer from acute pain.

In the current study the investigators will use a multistage approach to test the hypothesis whether the use of a CDSS in prehospital emergency care will: 1. Improve protocol adherence, 2. Reduce emergency department length of stay, 3. Improves diagnostic accuracy; without impeding the workflow of the prehospital team or impairing patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive treatment from the Paramedic Intervention Team (PIT) in the prehospital Emergency Medical Services (EMS) area of the University Hospitals, Leuven.

Exclusion Criteria:

* Patient-related interventions not dispatched by the Emergency Medical Dispatch center (EMD)
* Patient related interventions during transport between two healthcare facilities or in mass casualty situations.

Ages: 1 Year to 112 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Treatment protocol adherence | Up to 12 months
  Measured by comparing the prescribed actions to be taken following the selected standing order (-s) or procedures, with the actual action (-s) taken.

SECONDARY OUTCOMES:
Length of Stay in the ED | Up to 12 months
  Measured as the duration between the times the patient is assigned with a unique EAD number in the emergency department and the disposition decision is marked in the Electronic Patient Record (EPR), indicating that the patient is ready to be discharged from the ED.
Prehospital Patient Time Interval | Up to 12 months
  Measured as the duration between the arrival time at the scene and and arrival time at the ED.
Consistency in reported diagnose and the choice of PIT standing order (-s) or procedure (-s) | Up to 12 months
  Measured by comparing the selected standing order (-s) or protocol (-s) and the reported diagnose (-s).
Alignment between diagnostic accuracy and interventions taken. | Up to 12 months
  Measures by comparing the use of available scales and the corresponding prescribed action (-s) to be taken following the standing orders.

CONTACTS AND LOCATIONS:
Overall Officials: Bert mr Aertgeerts, PhD, Study Chair — Academic Center for General Practice
Locations (1):
- Academic Center for General Practice, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PhD Project — https://www.kuleuven.be/wieiswie/nl/person/00096106
- See also: Principal Investigator — http://goo.gl/i5mv0R
- See also: Participating Facility — http://goo.gl/sz9yDC
- See also: Affiliated study Department — http://goo.gl/UokRfN